CLINICAL TRIAL: NCT05654688
Title: GRASTON VERSUS MUSCLE ENERGY TECHNIQUE IN NONSPECIFIC NECK PAIN
Brief Title: NONSPECIFIC NECK PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Elsayed, Fellow of physical therapy Helwan University hospital, Egypt, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HelwanU
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Non Specific Neck Pain
Keywords: GRASTON TECHNIQUE

STUDY DESIGN:
Intervention Model Description: .Design: A randomized controlled experimental pre-post measurement. This study included forty two (30 males and 12 females) patients with NSNP aged between the ages of 40 and 60. Each participant was assigned a unique number, and then those numbers were randomly divided into three groups. Three groups were formed from a random selection of participants: GT Group (A): received 12 sessions of GT and (TPT) over the course of four weeks (three sessions per week). MET Group (B): received 12 sessions of MET treatment and (TPT) over a period of four weeks (three sessions per week). Control Group (C): received 12 sessions of traditional physiotherapy (TPT) over a period of four weeks (three sessions per week).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Graston (Experimental): Graston technique and traditional physical treatment (control)
  Interventions: Other: graston and muscle energy technique
- Muscle energy technique (Experimental): Muscle energy technique and traditional physical treatment
  Interventions: Other: graston and muscle energy technique
- Traditional physical therapy (Active Comparator): Traditional physical therapy treatment as heat application
  Interventions: Other: graston and muscle energy technique

INTERVENTIONS:
Other: graston and muscle energy technique — Graston technique (Gt) is a technique of mobilization of soft tissue using instruments which consider myofascial release instrument that has been reported to relieve pain, improve overall function, and increase range of motion.
  Muscle energy technique (MET) is a term composed of various types of active muscular relaxation and stretching procedures. The two cornerstone forms of MET are reciprocal inhibition and post isometric relaxation. In theory, reciprocal inhibition takes advantage of the neurological phenomena of muscular contraction, which results in an inhibitory effect on the antagonistic muscles.

SUMMARY:
The goal of this a randomized control trial is to carried out to examine Graston technique (GT) and muscle energy method (MET) impact on nonspecific neck pain compared to traditional physiotherapy treatment (TPT), This study aims to contrast between the outcomes of GT and MET on both pain intensity and functional disability in patients. Each participant was assigned a unique number, and then those numbers were randomly divided into three groups. Three groups were formed from a random selection of participants: GT Group (A): received 12 sessions of GT and (TPT) over the course of four weeks (three sessions per week). MET Group (B): received 12 sessions of MET treatment and (TPT) over a period of four weeks (three sessions per week). Control Group (C): received 12 sessions of traditional physiotherapy (TPT) over a period of four weeks (three sessions per week).

DETAILED DESCRIPTION:
Pain intensity (VAS) It was utilized to evaluate the degree of pain both before and after treatment. Subjects were asked to rate their pain on a scale from 0 (no pain) to 10 (extreme pain). Specifically, a line representing 10 centimeters was used as the scale's visual representation. Distance from zero to the respondent's mark was then used to approximate the sufferer's level of discomfort.

Functional Disability (NDI) The Neck Disability Index (NDI) is a 10-item questionnaire used to assess the functional impairment caused by neck pain. The questionnaire covers a wide range of topics related to one's everyday life, including but not limited to: personal care, heavy lifting, work, driving, sleeping, playing, recreational, pain level, concentration, and headache. Scores range from 0 (no disability) to 5 (severe disability) for each question, with the total score out of 100 determined by adding and doubling the scores for each question. If a patient has a high NDI score, they report being more disabled as a result of their neck pain. Patients have identified a 5-10% improvement as the "minimally clinically meaningful change." This study excluded any patient with: Symptoms or signs of upper motor neuron disease, vestibulobasilar insufficiency, and amyotrophic lateral sclerosis. Cervical spine fracture, Cases of disc prolapse that have been diagnosed (27), prior cervical or thoracic spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* non specific neck pain

Exclusion Criteria:

* Symptoms or signs of upper motor neuron disease, vestibulobasilar insufficiency, and amyotrophic lateral sclerosis.

Cervical spine fracture. Cases of disc prolapse that have been diagnosed. prior cervical or thoracic spine surgery, (28).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity (VAS) | 1 month
  Pain intensity (VAS) It was utilized to evaluate the degree of pain both before and after treatment. Subjects were asked to rate their pain on a scale from 0 (no pain) to 10 (extreme pain). Specifically, a line representing 10 centimeters was used as the scale's visual representation. Distance from zero to the respondent's mark was then used to approximate the sufferer's level of discomfort

SECONDARY OUTCOMES:
Functional Disability (NDI) | 1 month
  Functional Disability (NDI) The Neck Disability Index (NDI) is a 10-item questionnaire used to assess the functional impairment caused by neck pain. The questionnaire covers a wide range of topics related to one's everyday life, including but not limited to: personal care, heavy lifting, work, driving, sleeping, playing, recreational, pain level, concentration, and headache. Scores range from 0 (no disability) to 5 (severe disability) for each question, with the total score out of 100 determined by adding and doubling the scores for each question. If a patient has a high NDI score, they report being more disabled as a result of their neck pain. Patients have identified a 5-10% improvement as the "minimally clinically meaningful change."

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCormack JR, Underwood FB, Slaven EJ, Cappaert TA. Eccentric Exercise Versus Eccentric Exercise and Soft Tissue Treatment (Astym) in the Management of Insertional Achilles Tendinopathy. Sports Health. 2016 May/Jun;8(3):230-237. doi: 10.1177/1941738116631498. PMID 26893309